CLINICAL TRIAL: NCT06899880
Title: Perfusion Parameters and Outcome During a Standardized Deresuscitation Strategy with Net Ultrafiltration: a Retrospective Cohort Study.
Acronym: DeepCART
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 24-5563
Record Dates: First submitted 2025-03-21; First posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Fluid Overload; Acute Kidney Injury; Continuous Renal Replacement Therapy
MeSH Terms: conditions — Edema; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (1):
- Standardized deresuscitation strategy: Eligible patients without hypoperfusion benefited from: 1) a restrictive approach of intakes combining hypercaloric enteral or per os feeding with hydric restriction as much as possible and no fluid of maintenance, and 2) a systematic UFnet of 2 mL/kg/h until reaching dry weight and a systematic monitoring every 6 h of: peripheral perfusion by capillary refilling time and mottling score, arterial lactate level, and central venous oxygen saturation.
  Interventions: Other: Describe the perfusion parameters during a deresuscitation strategy and their association with the outcome.

INTERVENTIONS:
Other: Describe the perfusion parameters during a deresuscitation strategy and their association with the outcome. — Arterial lactate, pCO2 gap, SvO2, capillary refill time and mottling score anomalies will be described during the first 5 days of the deresuscitation strategy.

SUMMARY:
Hemodynamic tolerance of fluid removal during deresuscitation is a cornerstone of the impact on outcome of such a strategy. However, how to define and to predict hemodynamic tolerance to fluid removal remains controversial. The investigators routinely use a standardized deresuscitation protocol in patients with fluid overload and continuous renal replacement therapy combined with monitoring of clinical and biological perfusion parameters.

The aim of the study was to describe perfusion during deresuscitation, and to determine whether it is associated with major adverse kidney events at day 30.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Acute kidney injury requiring continuous renal replacement therapy
* Standardized deresuscitation following a routine care protocol

Exclusion Criteria:

* Chronic hemodialysis
* Advanced directives to withhold or withdraw life-sustaining treatment,
* Patient's opposition to the use of his/her personal health data

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: adults' patients with fluid overload and continuous renal replacement therapy in intensive care unit
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
MAKE 30 | A day 30 after the initiation of the deresuscitation strategy
  Major adverse kidney event at day 30, defined as follows:
  * Death OR
  * No weaning of renal replacement therapy OR
  * Serum creatinine > 2 times baseline serum creatinine

CONTACTS AND LOCATIONS:
Locations (1):
- Louis Pradel Hospital, France, Bron, France